CLINICAL TRIAL: NCT07343856
Title: Development of a Personalized Alternative Non-invasive Rapid Diagnostic Test for SARS-CoV-2 in Patients With Long COVID
Brief Title: Long COVID Diagnostic Reactivity Assesment Test
Acronym: EAV-LONGCOVID
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oncology Center,Ministry Of Heath,Uzbekistan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9/36-2216
Record Dates: First submitted 2025-12-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Long COVID; Post-Acute Sequelae of SARS-CoV-2 Infection
Keywords: Long COVID; Post-acute sequelae of SARS-CoV-2 infection; Bioelectrical assessment; Electroacupuncture diagnostics; Medicament testing; Autonomic dysregulation; Chronic viral persistence; Non-invasive diagnostics
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: All enrolled participants undergo a single-session diagnostic assessment using medicament testing to evaluate bioelectrical response patterns associated with viral persistence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic Assesment Arm (Experimental): This single-arm study includes participants undergoing a non-invasive electrodiagnostic assessment to evaluate bioelectrical response patterns associated with viral antigen persistence. No therapeutic intervention is administered.
  Interventions: Diagnostic Test: Electrodiagnostic Bioelectrical Assessment

INTERVENTIONS:
Diagnostic Test: Electrodiagnostic Bioelectrical Assessment — A non-invasive diagnostic procedure performed during a single session to assess bioelectrical response patterns associated with viral antigen persistence. Measurements are obtained using standardized bioelectrical assessment techniques without administration of any therapeutic agents or interventions.

SUMMARY:
This study is a diagnostic clinical investigation designed to evaluate bioelectrical response patterns assessed by electro-acupuncture-based medicament testing.

The method is used to identify individual bioelectrical reactivity associated with the presence and persistence of pathological factors and to assess patient-specific responses to tested medicinal substances.

The study involves a single-session, non-invasive diagnostic procedure without administration of pharmacological treatment. The primary objective is the methodological evaluation of the diagnostic approach and the characterization of the detected bioelectrical response patterns in the studied population.

DETAILED DESCRIPTION:
This study is a diagnostic clinical investigation designed to evaluate bioelectrical response patterns assessed by electro-acupuncture-based medicament testing.

The method is used to identify individual bioelectrical reactivity associated with the presence and persistence of pathological factors and to assess patient-specific responses to tested medicinal substances.

The study involves a single-session, non-invasive diagnostic procedure without pharmacological treatment. The primary objective is the methodological evaluation of the diagnostic approach and the characterization of the detected bioelectrical response patterns in the studied population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of confirmed SARS-CoV-2 infection
* Persistent symptoms consistent with Long COVID lasting ≥12 weeks after acute infection
* Ability to provide informed consent
* Willingness to undergo non-invasive bioelectrical diagnostic assessment

Exclusion Criteria:

* Acute infectious disease at the time of enrollment
* Severe uncontrolled medical or psychiatric conditions that may interfere with diagnostic assessment
* Implanted electronic medical devices (e.g., pacemaker)
* Pregnancy or breastfeeding
* Inability to comply with study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Bioelectrical Response Patterns Consistent With Viral Persistence | At enrollment (single diagnostic session)
  Non-invasive diagnostic assessment using electroacupuncture-based medicament testing to identify bioelectrical response patterns consistent with viral antigen persistence in participants with post-viral conditions.

SECONDARY OUTCOMES:
Distribution of Bioelectrical Reactivity Patterns During Medicament Testing | Baseline(Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Naylya Djumaeva, MD,PhD, Principal Investigator — Reseacrh Institute of Virology
Locations (1):
- Research Institute of Virology, Tashkent, Uzbekistan